CLINICAL TRIAL: NCT00129038
Title: A Randomised, Crossover Study Comparing the Biochemical and Platelet Effects of Modified-release Dipyridamole/Aspirin (200mg/25 mg bd; Asasantin Retard®) With Aspirin (75 mg qd) in Coronary Artery Disease Patients With Aspirin Resistance Manifesting as Persistent Thromboxane Formation.
Brief Title: Modified-release Dipyridamole/Aspirin (200mg/25mg bd) Versus Aspirin (75mg) in Aspirin-resistant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 9.169
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin

INTERVENTIONS:
Drug: modified-release dipyridamole/aspirin
Drug: aspirin

SUMMARY:
The primary objective of this study is to assess whether adding modified-release dipyridamole to aspirin (Asasantin Retard) has measurable effects on markers of platelet function (for example, platelet aggregation) in patients with cardiovascular disease who are known to be resistant to aspirin alone

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular disease (including history of stroke or transient ischaemic attack)
* Documented evidence of resistance to aspirin
* Capable of comprehending and communicating effectively with the investigator and staff and of providing informed consent.
* Willing to give informed consent prior to participation in the trial.

Exclusion Criteria:

* Any clinically significant condition other than cardiovascular disease.
* Clinically significant abnormal baseline haematology, blood chemistry or urinalysis findings.
* Use of dipyridamole, clopidogrel, ticlopidine or any non-steroidal anti-inflammatory agent (NSAID)(including COX-2 inhibitors) during the two weeks before randomisation and during the trial.
* Active peptic ulceration or history of peptic ulcer disease.
* Known history of or suspected hypersensitivity to dipyridamole, aspirin, any NSAID or any other component of the test drugs.
* History of any bleeding disorder.
* History of cerebral haemorrhage.
* Resting seated blood pressure less than 90/60mmHg.
* Participation in any drug clinical trial within sixteen weeks prior to the start of the trial.
* Any indication of current or previous abuse of alcohol, solvents or drugs.
* Asthma.
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (e.g. oral contraceptives, intrauterine devices or surgically sterile).
* Previous participation in the randomisation phase of this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2007-01-01 (Actual)

PRIMARY OUTCOMES:
platelet aggregation in response to arachidonic acid | baseline, day 14, day 30 of each period

SECONDARY OUTCOMES:
platelet aggregation in response to epinephrine, adenosine diphosphate (ADP) and collagen | baseline, day 14, day 30 of each period
serum thromboxane B2 | baseline, day 14, day 30 of each period
urinary 2,3,-dinor-6-keto-prostaglandin F1α | baseline, day 30 of each period
urinary 11-dehydro-thromboxane B2 | baseline, day 30 of each period
plasma CD40L | baseline, day 14, day 30 of each period
flow cytometry measurements of platelet receptors in blood samples | baseline, day 14, day 30 of each period
bleeding time | day 30 of each period
6-keto-prostaglandin F1α (in bleeding time samples) | day 30 of each period
thromboxane B2 (in bleeding time samples) | day 30 of each period
flow cytometry measurements from bleeding time samples | day 30 of each period]
coagulation markers F1.2 and fibrinopeptide A (in bleeding time samples) | day 30 of each period
pulse rate and blood pressure | baseline, day 14, day 30 of each period

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Ireland (2):
  - 9.169.01 Dept of Clinical Pharmacology, Dublin
  - 9.169.02 St. James' Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency